CLINICAL TRIAL: NCT03189576
Title: Measuring Molecular Residual Disease in Colorectal Cancer After Primary Surgery and Resection of Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Pirkko-Liisa Kellokumpu-Lehtinen, professor, Tampere University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ETL R15085
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Residual Disease
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm, Residual | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRC patients after primary surgery (Other): sequential blood draw taken to monitor residual disease
  Interventions: Diagnostic Test: blood draw

INTERVENTIONS:
Diagnostic Test: blood draw

SUMMARY:
Circulating tumour DNA (ctDNA) is a promising tool when monitoring the residual disease in colorectal cancer (CRC). Current staging procedures are insufficient to identify the patient cohort at high risk, who might benefit from additional adjuvant therapy.

We will show that the assessment of ctDNA is a non-invasive approach and easily taken at different time points via simple blood draw to monitor residual disease from the colorectal cancer patients after primary surgery. Minimal residual disease could be used in the future for individualized treatment decisions after primary surgery.

ELIGIBILITY:
Inclusion Criteria:

* planned colorectal primary surgery

Exclusion Criteria:

* unfit patients with dementia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
ctDNA level | 3-6 months
  residual disease measured by sequential blood draws

CONTACTS AND LOCATIONS:
Overall Officials: Pirkko-Liisa Kellokumpu-Lehtinen, professor, Study Director — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No